CLINICAL TRIAL: NCT03743740
Title: The Effect of Spinal Stabilization Exercises on Fatigue, Muscle Strength, Pulmonary Functions and Functional Capacity in Patients With Myasthenia Gravis
Brief Title: The Effect of Spinal Stabilization Exercises in Patients With Myasthenia Gravis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ali Naim Ceren, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KA-17132
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): first, patients will undergo spinal stabilization exercise and home based program 3 days per week for 6 weeks.
  then, exercises will be suspended for 4 weeks. then, patients will undergo home based program 3 days per week for 6 weeks.
  Interventions: Other: Spinal stabilization exercise
- Group 2 (Experimental): first, patients will undergo home based program 3 days per week for 6 weeks. then, exercises will be suspended for 4 weeks. then, patients will undergo spinal stabilization exercise and home based program 3 days per week for 6 weeks.
  Interventions: Other: Spinal stabilization exercise

INTERVENTIONS:
Other: Spinal stabilization exercise — The effects of spinal stabilization exercise in patients with myasthenia gravis will be investigated.There is no study in the literature that previously applied spinal stabilization exercises in patients with myasthenia gravis. The benefits of spinal stabilization exercises in other diseases are shown.
  Other Names: home based program

SUMMARY:
Myasthenia Gravis (MG) is an autoimmune disease characterized by increased exercise-induced fatigue and muscle weakness. MG is a disease caused by impaired receptor function due to antibodies to nicotinic acetylcholine receptors in postsynaptic region in voluntary skeletal muscles.Spinal stabilization exercises, which use the basic principles of motor learning, aiming to improve the coordination, contraction rate and endurance of the body muscles by increasing kinesthetic awareness, can be used to strengthen body stability.

The aim of this study was to investigate the effects of spinal stabilization exercises on fatigue, muscle strength, pulmonary functions and functional capacity in patients with MG.

DETAILED DESCRIPTION:
Myasthenia Gravis (MG) is an autoimmune disease characterized by increased exercise-induced fatigue and muscle weakness. MG is a disease caused by impaired receptor function due to antibodies to nicotinic acetylcholine receptors in postsynaptic region in voluntary skeletal muscles. The disease usually begins with ptosis from ocular symptoms. With the progression of the disease, symptoms of bulbar muscles and extremity muscles are added to the ocular symptoms. Bulbar symptoms occur when speaking, swallowing, chewing difficulties and difficulty breathing, while the symptoms in the extremity muscles arise as the difficulty of raising the arms uphill and the strain of climbing stairs.

The weakness of the limb muscles is proximal and distal in the arms and more proximal muscles in the legs. As the disease progresses, weakness occurs in most striated muscles. This causes weakness in the trunk muscles.

In the literature, the physiotherapy methods used in MG patients include breathing exercises, aerobic exercises and resistant exercises.Spinal stabilization exercises enable activation of the trunk muscles.

Spinal stabilization exercises, which use the basic principles of motor learning, aiming to improve the coordination, contraction rate and endurance of the body muscles by increasing kinesthetic awareness, can be used to strengthen body stability. Spinal stabilization exercises are a type of exercise that aims more smooth limb movements with a strong spine, ensuring smoothness and stability of the spine. In the literature, there is no study using spinal stabilization exercises in MG patients. The aim of this study was to investigate the effects of spinal stabilization exercises on fatigue, muscle strength, pulmonary functions and functional capacity in patients with MG.

Method The study was planned as randomized, single-blind and cross-over. Randomization will be done with closed envelope system. Group 1 will be written on five sheets and group 2 will be written on another five sheets.

Then, these papers will be placed on the envelopes, these envelopes will be mixed in a box and patients will be asked to withdraw from these envelopes.

Thus, patients will be divided into 2 groups. Assessments will be made by Yeliz Salcı and Ebru Kütük Çalıkçı. The assessors will not know who is in the which group. Treatment intervention will be done by Ali Naim Ceren. The assessors will evaluate patients without knowing the patients' groups. So the work will be single blind. Group 1, 3 days per week for 6 weeks so that it will be taken to the physiotherapy program consisting of spinal stabilization exercises. Also the treatment will be supported by home program exercises. The patients will be rested for 4 weeks to eliminate the effects of the spinal stabilization program. After this period, only the home program will be given for 6 weeks. In Group 2; treatment will start with a 6-week home program, followed by a 4-week break.

At the end of this period to be 3 days a week for 6 weeks spinal stabilization exercise program will be implemented. In addition to this exercise program, patients will be given a home program. The home program will include breathing exercises tailored to the patient's needs, calisthenic exercises, and MAT activities.

Assessments will be made at the beginning of the treatment, after 6 weeks of treatment, at the end of 4 weeks of rest and at the end of 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MG by a neurologist,
* Aged between18-65 years,
* To be in Stage II or III according to the Clinical Classification of the Medialia Gravis Functional Assessment (MGFA),
* The Mini Mental Test score should be over 24 in order to be cooperative to the physiotherapist's instructions,
* To volunteer to participate in the study.

Exclusion Criteria:

* Having a cognitive problem and having a Mini Mental Test score below 24
* To have had myasthenic crisis in the last month,
* Modification of medical treatment and dose in the last month,
* Systemic, orthopedic and neurological disease in addition to the disease
* Participation in physiotherapy program in the last six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
muscle strength of extremity muscle in patient with Myasthenia Gravis | 6 weeks
  change in muscle strength will be measured with a digital hand held dynamometer
fatigue perception | 6 weeks
  fatigue perception will be assessed with visual analog scale (VAS). VAS is a straight line with a length of 10 cm meaning of 0 is that I am not tired. The meaning of 10 is that I am too tired. According to the degree of fatigue patients feel, patients give a score in this range.
fatigue | 6 weeks
  fatigue will be assessed with fatigue severity scale (FSS). FSS is a scale with scores ranging from 7 to 63. It includes 9 questions. Increase of score in this scale means that fatigue severity is increasing.
respiratory functions | 6 weeks
  respiratory functions will be assessed with respiratory function tests. Respiratory function tests will be performed with portable spirometry.
functional capacity | 6 weeks
  functional capacity will be assessed with 6 minute walk test. The 6-minute walk test will record the distance traveled in the 30-meter corridor at maximal speed for 6 minutes.

SECONDARY OUTCOMES:
Quality of Life Assessment | 6 weeks
  It will be evaluated with Myastenia GravisvQuality of Life Questionnaire 15

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gilhus NE. Myasthenia Gravis. N Engl J Med. 2016 Dec 29;375(26):2570-2581. doi: 10.1056/NEJMra1602678. No abstract available. PMID 28029925
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Background] Nicolle MW. Myasthenia Gravis and Lambert-Eaton Myasthenic Syndrome. Continuum (Minneap Minn). 2016 Dec;22(6, Muscle and Neuromuscular Junction Disorders):1978-2005. doi: 10.1212/CON.0000000000000415. PMID 27922503
- [Background] Feasson L, Camdessanche JP, El Mandhi L, Calmels P, Millet GY. Fatigue and neuromuscular diseases. Ann Readapt Med Phys. 2006 Jul;49(6):289-300, 375-84. doi: 10.1016/j.annrmp.2006.04.015. Epub 2006 Apr 25. English, French. PMID 16780988
- [Background] Elsheikh B, Arnold WD, Gharibshahi S, Reynolds J, Freimer M, Kissel JT. Correlation of single-breath count test and neck flexor muscle strength with spirometry in myasthenia gravis. Muscle Nerve. 2016 Jan;53(1):134-6. doi: 10.1002/mus.24929. PMID 26437790
- [Background] Salci Y, Karanfil E, Balkan AF, Kutukcu EC, Ceren AN, Ayvat F, Bekircan-Kurt CE, Armutlu K. Functional exercise capacity evaluated by timed walk tests in myasthenia gravis. Muscle Nerve. 2019 Feb;59(2):208-212. doi: 10.1002/mus.26345. Epub 2018 Oct 17. PMID 30230561
- [Background] Yang Y, Zhang M, Guo J, Ma S, Fan L, Wang X, Li C, Guo P, Wang J, Li H, Li Z. Quality of life in 188 patients with myasthenia gravis in China. Int J Neurosci. 2016;126(5):455-62. doi: 10.3109/00207454.2015.1038712. Epub 2015 Jun 5. PMID 26000922